CLINICAL TRIAL: NCT00813098
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Determine the Safety and Efficacy of Orally Administered LX1031 in Subjects With Non-Constipating Irritable Bowel Syndrome
Brief Title: Study of LX1031 in Subjects With Non-Constipating Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Joel P. Freiman, MD, MPH / Medical Director Drug Safety, Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol LX1031.1-201-IBS; LX1031.201 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — 2-amino-3-(4-(2-amino-6-(2,2,2-trifluoro-1-(3'-methoxybiphenyl-4-yl)ethoxy)-pyrimidin-4-yl)phenyl)propionic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose (Experimental): A high dose of LX1031; daily oral intake for 28 days
  Interventions: Drug: LX1031 High Dose
- Low Dose (Experimental): A low dose of LX1031; daily oral intake for 28 days
  Interventions: Drug: LX1031 Low Dose
- Placebo (Placebo Comparator): Matching placebo dosing with daily oral intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LX1031 High Dose — A high dose of LX1031; daily oral intake for 28 days
  Arms: High dose
Drug: LX1031 Low Dose — A low dose of LX1031; daily oral intake for 28 days.
  Arms: Low Dose
Drug: Placebo — Matching placebo dosing with daily oral intake
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and effectiveness of LX1031 versus a placebo control in subjects with non-constipating irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-70 years old
* Documented diagnosis of IBS (IBS-diarrhea or IBS-mixed) based upon Rome III criteria
* Abdominal pain/discomfort at least 2 days per week during the screening and run-in periods
* Normal structural evaluation of the colon within 5 years prior to screening
* Ability to provide written informed consent

Exclusion Criteria:

* Inability to discontinue current drug therapy for IBS, except for bulking agents, through the duration of the study
* Use of anticholinergic antidepressants, opioid pain medications, or any drugs that affect bowel motility
* Lactose intolerance
* Major psychological disorder
* Significant nicotine or caffeine use (>10 cigarettes and/or six 8 ounce cups of coffee per day, respectively)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel P. Freiman, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (36):
- United States (36):
  - Genova Clinical Research, Tucson, Arizona
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Edinger Medical Group Clinical Research Center, Fountain Valley, California
  - Impact Clinical Trials, Los Angeles, California
  - Community Clinical Trials, Orange, California
  - AGMG - Orange, Orange, California
  - Medical Associates Research Group, San Diego, California
  - Lynn Instiute of the Rockies, Colorado Springs, Colorado
  - Clinical Trials Management of Boca Raton, Inc., Boca Raton, Florida
  - Consultants for Clinical Research of S. Florida, Boynton Beach, Florida
  - Research Consultants Group, Hialeah, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - ActivMed Practice and Research, Haverhill, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Long Island Clinical Research, Great Neck, New York
  - Cary Medical Research, Cary, North Carolina
  - The UNC Center for Functional GI & Motility Disorders, Chapel Hill, North Carolina
  - Medoff Medical/Vital re:Search, Greensboro, North Carolina
  - Unifour Medical Research, Hickory, North Carolina
  - Piedmont Medical Associates, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Gastroenterology Research Consultant of Greater Cincinnati, Cincinnati, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Coastal Carolina Research Center in Goose Creek, Goose Creek, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Pioneer Research Solutions, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Advanced Research Institute, Ogden, Utah
  - Utah Clinical Trials, LLC, Salt Lake City, Utah
  - National Clinical Research Norfolk Inc., Norfolk, Virginia
  - Aurora Health Center - Waukesha, Waukesha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center trial in the United States, with 36 investigators participating.
Pre-assignment Details: There was a 14-day Run-in period before randomization.
Period: Overall Study
Arm/Group | High Dose | Low Dose | Placebo
Started | 49 | 54 | 52
Completed | 46 | 46 | 50
Not Completed | 3 | 8 | 2
Not completed — Adverse Event | 2 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Inability to complete study procedures | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Principal Investigator decision | 0 | 1 | 0
Not completed — Withdrew Consent | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Placebo | Total
Number analyzed (Participants) | 43 | 44 | 47 | 134
Age Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.24) | 46.7 (13.34) | 48.0 (12.70) | 47.8 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants] — Measure based upon the per protocol population
  Participants
    Female | 34 | 36 | 7 | 77
    Male | 9 | 8 | 40 | 57
Race/Ethnicity, Customized [Number; unit: participants] — Measure based upon the per protocol population.
  participants
    White | 37 | 40 | 44 | 121
    Black or African American | 6 | 3 | 1 | 10
    Asian | 0 | 0 | 1 | 1
    Other | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 47 | 134
IB Sub-type [Number; unit: participant] — Measure based upon the per protocol population. Non-constipating IBS patients entering the trial were classified into 2 groups: irritable bowel syndrome-diarrhea (IBS-D) or irritable bowel syndrome-mixed (IBS-M).
  participant
    IBS-M | 9 | 9 | 12 | 30
    IBS-D | 34 | 35 | 35 | 104

OUTCOME MEASURES:

1. Primary Outcome: Subjects Who Experienced Relief of IBS Pain and Discomfort at Week 4
Description: The primary efficacy endpoint was the proportion of subjects experiencing relief of IBS pain and discomfort at Week 4 as measured by the response to the question,"In the past 7 days have you had adequate relief of your irritable bowel syndrome pain and discomfort?"
Time Frame: Week 4
Population: Per protocol population; Last observation carried forward.
Measure: Number; unit: Participants
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 43 | 44 | 47
Participants | 23 | 18 | 20

2. Secondary Outcome: Change From Baseline at Week 4 in Proportion of Days Per Week When Experiencing Urgency to Defecate
Description: To assess sensation of urgency to defecate on a daily basis, subjects recorded in their daily diary a response to the following question,"Have you felt or experienced a sense of urgency to pass stool today?" The mean score (proportion of days per week when the subject experienced an urge to defecate) for Week 4 was subtracted from the baseline mean score to determine the mean change from baseline.
Time Frame: Baseline to Week 4
Population: Per protocol population; Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 43 | 44 | 47
Score on a scale | -0.32 (0.367) | -0.26 (0.252) | -0.33 (0.369)

3. Secondary Outcome: Change From Baseline at Week 4 in Stool Consistency Scores
Description: Stool consistency was evaluated using the 7-point Bristol Stool Scale in which a score of 1 indicates separate hard lumps, 2 indicates sausage shaped but lumpy, 3 indicates sausage-like with cracks on the surface, 4 indicates sausage-like but smooth and soft, 5 indicates soft blobs with clear cut edges, 6 indicates fluffy pieces with ragged edges, and 7 indicates watery with no solid pieces. The mean score for Week 4 was subtracted from the baseline mean score to obtain the mean change from baseline.
Time Frame: Baseline to Week 4
Population: Per protocol population; Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 43 | 44 | 47
Score on a scale | -1.11 (0.920) | -0.30 (0.877) | -0.56 (1.187)

4. Secondary Outcome: Change From Baseline at Week 4 in Stool Frequency
Description: Subjects recorded the number of times they passed stool on a daily basis in the daily diary. The mean for Week 4 was subtracted from the baseline mean to obtain the mean change from baseline in stool frequency.
Time Frame: Baseline to Week 4
Population: Per protocol population; Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Number of daily stools
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 43 | 44 | 47
Number of daily stools | -0.75 (1.021) | -0.52 (0.921) | -0.62 (0.970)

5. Secondary Outcome: Change From Baseline at Week 4 on the Severity of Bloating
Description: Subjects recorded in the daily diary the level of bloating they felt on a daily basis using a 100 mm visual analog scale (with 0 being "not at all" and 100 mm being "worst possible"). The mean score for Week 4 was subtracted from the baseline mean score to obtain the mean change from baseline in severity of bloating.
Time Frame: Baseline to Week 4
Population: Per protocol population; Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 43 | 44 | 47
Score on a scale | -18.68 (20.922) | -15.13 (15.469) | -15.48 (25.855)

6. Secondary Outcome: Change From Baseline at Week 4 on the Global Improvement Score.
Description: The IBS Global Improvement Scale (IBS-GAI) asks "Compared to the way you felt before you entered the study, have your IBS symptoms over the past 7 days been: 1-substantially worse, 2-moderately worse, 3-slightly worse, 4-no change, 5-slightly improved, 6-moderately improved, 7-substantially improved?" The mean score for Week 4 was subtracted from the mean baseline score to obtain the mean change from baseline on the Global Improvement Score.
Time Frame: Baseline to Week 4
Population: Per protocol population; Last observation carried forward.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose | Low Dose | Placebo
Number analyzed (Participants) | 43 | 44 | 47
Score on a scale | 1.56 (1.501) | 1.33 (1.459) | 1.47 (1.666)

ADVERSE EVENTS:
Time Frame: Adverse events were followed at the start of study drug to no more than 14 days (30 days for serious adverse events) after the last dose of study drug.
Arm/Group | High Dose | Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 11/49 | 11/54 | 13/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=49) | Low Dose (N=54) | Placebo (N=52)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=49) | Low Dose (N=54) | Placebo (N=52)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (6)
Nausea (Gastrointestinal disorders) | 4 (12) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 1 (2) | 2 (3)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that written permission be given before the PI can release any data publicly.